CLINICAL TRIAL: NCT04696146
Title: A Phase I/II, Double-Blind, Placebo-Controlled Study: Assessing Safety and Efficacy of Preoperative Renal Allograft Infusions of C1 Inhibitor (Berinert®) (Human) (C1INH) vs. Placebo Administration in Recipients of a Renal Allograft From Deceased High Risk Donors and Its Impact on Delayed Graft Function (DGF) and Ischemia/Reperfusion Injury (IRI)
Brief Title: Berinert (C1INH) vs Placebo for DGF/IRI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: OneLegacy Foundation (Unknown)
Responsible Party: Principal Investigator, Stanley Jordan, MD, Director of Nephrology and Transplant Immunology, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 469
Record Dates: First submitted 2020-12-22; First posted 2021-01-06 (Actual); Results first posted 2023-09-29 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: End Stage Renal Disease; Chronic Kidney Diseases
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — Complement C1 Inhibitor Protein; Saline Solution

STUDY DESIGN:
Intervention Model Description: Intraoperative C1INH (500U/kidney) vs. Placebo administered into the graft renal artery 1-2 hours prior to implantation in adult subjects receiving a deceased donor kidney allograft considered high-risk for development of DGF (KDPI>80). Patients will be randomized in a 1:1 manner
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Once eligible patients are identified, consented, and have an acceptable kidney transplant offer, they will be randomized by the Cedars-Sinai Research Pharmacy to receive study drug vs. placebo. Drug and placebo will be prepared by the Cedars-Sinai Research Pharmacy and conveyed to the operating room in a blinded manner. The drug will be administered by the transplant surgeon in the OR in a blinded manner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Berinert (Experimental): Berinert 500 units
  Interventions: Drug: Berinert
- Placebo (Placebo Comparator): Normal Saline in identical volume to Berinert
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Berinert — Intrarenal dose of 500 U of Berinert
  Other Names: C1 Esterase Inhibitor (C1INH)
  Arms: Berinert
Drug: Placebo — Normal Saline placebo
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
This is a Phase I/II double-blind, randomized, placebo-controlled study assessing safety and limited efficacy of intraoperative C1INH (500U/kidney) vs. Placebo administered into the graft renal artery 1-2 hours prior to implantation in adult subjects receiving a deceased donor kidney allograft considered high-risk for development of DGF (KDPI>80). Once eligible patients are identified, consented, and have an acceptable kidney transplant offer, they will be randomized by the Cedars-Sinai Research Pharmacy to receive study drug vs. placebo. Drug and placebo will be prepared by the Cedars-Sinai Research Pharmacy and conveyed to the operating room in a blinded manner. The drug will be administered by the transplant surgeon in the OR in a blinded manner.

DETAILED DESCRIPTION:
Pre-operative, infusion of C1INH into the renal allograft artery 1-2 hours prior to implantation will improve early graft function and reduce the rate of DGF, requirements for dialysis, graft survival and eGFR in patients receiving kidney allografts from high risk deceased donor compared to placebo.

Early graft function has a long-term effect on graft survival. Poor early graft function and DGF contributes to decreased short- and long-term patient and graft survival, increased incidence of acute rejection, prolonged hospitalization, and higher costs of transplantation. Although multiple factors contribute to the impaired graft function, ischemia-reperfusion injury (IRI) is the underlying pathophysiology leading to poor early graft function and DGF. A >35% incidence of DGF has remained constant over time despite significant improvements in immunosuppressive strategies and patient management. This may be due to increased use of kidneys from "extended-criteria" and/or non-heart-beating donors, where even greater rates (>60%) of DGF have been reported.

More than 94,653 people are currently waiting for a kidney transplant in the United States (UNOS.org 9/30/2019). Of the 19,360 kidney transplants performed in the US in 2018, 20% were from DCD donors and 9% from donors of KDPI>85. The USRDS reports that more than 50% of patients on the waiting list are willing to accept a kidney from an expanded-criteria donor (KDPI >85). This study will seek to expand the use of high KDPI kidneys and reduce wastage by showing improved function after C1INH treatment.

Patients who fulfill all I/E criteria will be eligible to be enrolled into Study

I Study Group (40 patients):

Treatment Arm I - KDPI >80 kidneys will be infused with one intrarenal dose of 500U of Berinert® in OR prior to implantation into the recipient.

Control Arm - KDPI >80 kidneys will be administered one intrarenal dose of normal saline (NS) in the OR in a volume identical to the volume of the dose of Berinert® before implantation of kidney into the patient.

Drug v. placebo administration will be randomized 1:1. Drug preparation and randomization will be carried out in a blinded fashion by research pharmacist.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men or women (18-70 years of age) who are on chronic dialysis therapy and acceptable candidates for receipt of a kidney transplant.
2. Recipients who are ABO compatible with donor allograft
3. Understand and sign a written inform consent prior to any study specific procedure
4. Women of childbearing potential must have a negative pregnancy test prior to randomization, and must be on an acceptable form of birth control.
5. . AND one of the below criteria:

   a)Recipients of kidney allograft from KDPI >80 donors b)Recipients of kidney allograft from DCD donors c)Recipients of kidney allograft with CIT > 24 hours d)Recipients of kidney allograft from donor on HD/CRRT prior to death/procurement e)Recipients of kidney allograft with donor terminal creatinine SCr ≥3.0 mg/dL f)Patient risk a total risk index score of >/=3

Exclusion Criteria:

1. Patients with a known pro-thrombotic disorder. (eg. Factor V Leiden)
2. Patients with a history of thrombosis or hypercoagulable state, excluding access clotting.
3. Patients with a history of administration of C1INH containing products or recombinant C1INH within 15 days prior to study entry.
4. Patients with a known hypersensitivity to treatment with C1INH.
5. Patients with an abnormal coagulation function. (INR>2, PTT> 50, PLT<60,000)who are not on anti-coagulation.
6. Patients with known active presence of malignancies.
7. Patients who arePCR positive for Hep B, Hep C, or HIV.
8. Recipients of pre-emptive kidney transplantation.
9. All zero mismatch kidneys.
10. Recipients of multi-organ transplants. (kidney and any other organ)
11. Recipients of kidney allograft that was on pump preservation for any period prior to transplantation.
12. Recipients of kidney allograft from a living donor.13)Female subjects who are pregnant or lactating.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Huang E, Ammerman N, Vo A, Hou J, Kumar S, Badash N, Falk B, Hernando K, Gillespie M, Kim IK, Lim K, Najjar R, Peng A, Shin B, Steggerda JA, Todo T, Brennan TV, Voidonikolas G, Wisel SA, Heeger PS, Jordan SC. Back-table intra-arterial administration of C1 esterase inhibitor to deceased donor kidney allografts improves posttransplant allograft function: Results of a randomized double-blind placebo-controlled clinical trial. Am J Transplant. 2025 Sep;25(9):1926-1939. doi: 10.1016/j.ajt.2025.05.003. Epub 2025 May 9. PMID 40349965

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Berinert | Placebo
Started | 21 | 24
Completed | 20 | 20
Not Completed | 1 | 4
Not completed — Transplant Cancelled and did not proceed with study | 0 | 4
Not completed — Off hours issue with product | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Berinert | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [53 to 64] | 63 [53 to 69] | 59 [53 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 4 | 17
  Male | 7 | 16 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 12 | 25
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Need for Dialysis in the First 30 Days Post-transplant
Description: The percentage of patients enrolled who require at least one session of dialysis in the first 30 days post transplant.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Berinert | Placebo
Number analyzed (Participants) | 20 | 20
Participants | 10 | 10

2. Primary Outcome: Renal Function 6 Months
Description: eGFR at 6M post-transplant
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ml/min/1.73m^2
Arm/Group | Berinert | Placebo
Number analyzed (Participants) | 20 | 20
ml/min/1.73m^2 | 54 (19) | 42 (14)

3. Primary Outcome: Graft Survival 6 Months
Description: Number of participants with graft survival at 6 Months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Berinert | Placebo
Number analyzed (Participants) | 20 | 20
Participants | 20 | 20

4. Secondary Outcome: Rejection Episodes at 6 Months
Description: Number of participants with a rejection episodes by day 180
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Berinert | Placebo
Number analyzed (Participants) | 20 | 20
Participants | 3 | 0

5. Secondary Outcome: Development of Donor Specific Antibodies (DSA) at 6 Months
Description: Number of participants with Donor Specific Antibodies (DSA) at 6 Months
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Berinert | Placebo
Number analyzed (Participants) | 20 | 20
Participants | 1 | 1

6. Other Pre Specified Outcome: Adverse Events in the Study Population
Description: Number of participants with an adverse events and serious adverse events
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Berinert | Placebo
Number analyzed (Participants) | 20 | 20
Participants | 16 | 17

ADVERSE EVENTS:
Time Frame: Adverse Event monitoring occurred from study enrollment to Day 180.
Arm/Group | Berinert | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 6/20 | 4/20
Other Adverse Events (participants affected / at risk) | 13/20 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Berinert (N=20) | Placebo (N=20)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Fever/sepsis (Infections and infestations) | 0 (0) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 2 (2)
Hyperkalemia (General disorders) | 0 (0) | 2 (3)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertensive urgency (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1)
Recurrent intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Generalized weakness (General disorders) | 0 (0) | 1 (1)
Partial small bowel obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0)
Visual disturbance (black spots), convulsions (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Berinert (N=20) | Placebo (N=20)
Hyperkalemia (General disorders) | 6 (6) | 11 (12)
Hyperglycemia (Endocrine disorders) | 5 (5) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT04696146/Prot_SAP_000.pdf